CLINICAL TRIAL: NCT04560582
Title: Immunosuppression Reduction in Failed Allograft Guided by cfDNA
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEPH-2018-27080
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant; Complications; Kidney Transplant Rejection; Kidney Transplant Failure
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be stored by study code. All study data will be associated with the specimen through the study code link.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney Transplant Patients with Failed Allograft: All participants are assigned to a single cohort of kidney transplant patients with failed allograft requiring dialysis.
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Participants will have blood drawn for analysis at baseline and every 4 weeks for a total of 7 blood draws over 24 weeks.

SUMMARY:
The optimal timing for immunosuppression tapering for patients with failed kidney transplant is not known. This pilot study would be to correlate rise in cf-DNA and increase in cPRA.

DETAILED DESCRIPTION:
This is an observational cohort study collecting data and blood specimens at designated time points. The primary outcome will be comparing the cPRA in patients that have a rise in cf-DNA to those that do not have a rise in cf-DNA. Seondary outcomes include comparison of the combined incidence of need for transfusion, need for methylprednisolone and allograft nephrectomy, ESA dose, allograft tenderness, and gross hematuria.

ELIGIBILITY:
Inclusion Criteria:

* Failed allograft requiring dialysis
* No living donor available for re-transplant option or anticipated deceased donor within the next 12 months
* Patient to be enrolled prior to 3rd HD (hemodialysis) session or within 1 week of starting peritoneal dialysis

Exclusion Criteria:

* 17 years or younger
* cPRA at entrance of 100%
* Primary non-function of the allograft
* Multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study proposes to recruit adult patients primarily from the inpatient units at UMMC Fairview, or the Renal or Transplant facilities at the Clinics and Surgery Center as attended by the PI and Co-Is. Additional clinics will be recruited from depending on patient population and clinician support.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
cPRA Concentrations | 1 day
  Outcome is reported as the serum concentration of calculated Panel Reactive Antibody (cPRA) at baseline.
cf-DNA Concentrations | up to 24 weeks
  Outcome is reported as the serum concentration of circulating-free DNA (cfDNA) at baseline, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks.

SECONDARY OUTCOMES:
Incidence of Need for Transfusion | 24 weeks
  Outcome is reported as the percent of participants who require transfusion.
Incidence of Need for Methylprednisolone and Allograft Nephrectomy | 24 weeks
  Outcome is reported as the percent of participants who require methylprednisolone and allograft nephrectomy
Incidence of ESA Dose | 24 weeks
  Outcome is reported as the percent of participants who require a erythropoesis stimulating agent (ESA) dose.
Incidence of Allograft Tenderness | 24 weeks
  Outcome is reported as the percent of participants who experience allograft tenderness.
Incidence of Gross Hematuria | 24 weeks
  Outcome is reported as the percent of participants who experience gross hematuria.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bregman, MD, Principal Investigator — University of Minenesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States